CLINICAL TRIAL: NCT05548777
Title: Andexanet Alfa and 4F-PCC Use in Patients Hospitalised With an Anticoagulant-related Major Bleed
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Outcomes Insights (Unknown)
Responsible Party: Sponsor
Other Study IDs: D9603R00004
Record Dates: First submitted 2022-08-26; First posted 2022-09-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Anticoagulant-related Major Bleed
MeSH Terms: interventions — PRT064445; Factor IX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients hospitalized for an anticoagulation-related major bleed
  Interventions: Drug: Andexanet alfa; Drug: 4F-PCC

INTERVENTIONS:
Drug: Andexanet alfa — Andexanet alfa
Drug: 4F-PCC — Four-Factor Prothrombin Complex Concentrate (4F-PCC)

SUMMARY:
This is an observational study based on data collected via an audit of electronic medical charts. The study population will include adult US patients treated with andexanet alfa or 4F-PCC during a hospitalization for an anticoagulation-related major bleed, and their characteristics, treatments and outcomes will be described.

DETAILED DESCRIPTION:
This observational study will include adult US patients treated with andexanet alfa or 4F-PCC during a hospitalization for an anticoagulation-related major bleed. Data will be collected via an audit of electronic medical charts. The primary objectives are to describe the patients' characteristics, treatments and outcomes, including length of stay and in-hospital mortality. Secondary objectives include subgroup analyses, including by bleed location. Potential differences between patients treated with andexanet alfa versus 4F-PCC, and potential differences in patient characteristics over time, will be assessed. If this assessment confirms that treatment groups can be adequately balanced and that patient characteristics have not substantially changed over time (i.e. no channeling bias is observed), the risk of in-hospital mortality with andexanet alfa versus 4F-PCC will be assessed in a comparative effectiveness analysis. If treatment groups cannot be balanced or clear signs of channelling bias are observed, the comparative analyses will be considered unfeasible and will not be performed.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10-CM diagnosis code of D68.32 (Hemorrhagic disorder due to extrinsic circulating anticoagulants) as part of an inpatient admission
* Taking either an oral FXa inhibitor or enoxaparin at the time of hospitalization for their bleeding event
* Treated with either andexanet alfa or 4F-PCC during the hospitalization for their bleeding event
* Had documented discharge disposition

Exclusion Criteria:

* Less than 18 years old
* Treated with both andexanet alfa and 4F-PCC during the hospitalization for their bleeding event

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult US patients treated with andexanet alfa or 4F-PCC during a hospitalization for an anticoagulation-related major bleed
Sampling Method: Probability Sample
Enrollment: 5480 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Mortality | During hospitalisation, approximately 6 days
  In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Agoura Hills, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AstraZeneca disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. AstraZeneca will accept request for IPD, but this does not mean requests will be granted and data shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: If and when a request has been approved, AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Dobesh PP, Coleman CI, Danese M, Lesen E, Chang RC, Odelade O, Fermann GJ. Management of factor Xa inhibitor-related traumatic non-intracranial bleeding events with andexanet alfa or four-factor prothrombin complex concentrate in a US multicenter observational study. J Am Coll Emerg Physicians Open. 2024 Nov 7;5(6):e13333. doi: 10.1002/emp2.13333. eCollection 2024 Dec. PMID 39524040
- [Derived] Dobesh PP, Fermann GJ, Christoph MJ, Koch B, Lesen E, Chen H, Lovelace B, Dettling T, Danese M, Ulloa J, Danese S, Coleman CI. Lower mortality with andexanet alfa vs 4-factor prothrombin complex concentrate for factor Xa inhibitor-related major bleeding in a U.S. hospital-based observational study. Res Pract Thromb Haemost. 2023 Aug 30;7(6):102192. doi: 10.1016/j.rpth.2023.102192. eCollection 2023 Aug. PMID 37753225
- See also: Redacted CSR synopsis_D9603R00004 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9603R00004&attachmentIdentifier=bfb47b8f-f18d-454a-a13a-11c9e45da538&fileName=CSR_synopsis_Acute_Major_Bleed_Chart_Audit_D9603R00004.pdf&versionIdentifier=